CLINICAL TRIAL: NCT00923156
Title: ESCAPE-SHF: A Double-blind, Double-dummy, Randomized, Multicenter, Parallel Group Study to Evaluate the Effects of Aliskiren, Ramipril and Combination Treatment on Plasma Concentration of Angiotensin II in Patients With Decompensated Systolic Heart Failure
Brief Title: Effects of Aliskiren, Ramipril, and the Combination on Levels of Angiotensin II in Patients With Decompensated Systolic Heart Failure
Acronym: ESCAPE-SHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100A2252; EudraCT 2008-001035-35
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-03-05 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Systolic; Aliskiren; Ramipril; Angiotensin II; Ang II; Plasma Renin Activity; PRA; Plasma Renin Concentration; PR,; brain natriuretic peptide; BNP; urinary aldosterone; Escape; Pharmacokinetic; PK
MeSH Terms: conditions — Heart Failure; Systolic Murmurs | interventions — aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Aliskiren (Experimental): In open label run-in phase (period 1), patients started with ramipril 2.5 mg or 5.0 mg capsule once daily (o.d) depending on previous treatment with RAAS blockers and up-titrated to ramipril 10 mg capsule o.d by end of period 1. In double blind phase (Period 2), patients received aliskiren (150 mg once daily) up titrated to 300 mg once daily after 1 week of treatment following a clinical safety patient assessment at the study site and matching placebo of ramipril capsules.
  Interventions: Drug: aliskiren; Drug: ramipril; Drug: Placebo to ramipril
- Ramipril (Experimental): In open label run-in phase (period 1), patients started with ramipril 2.5 mg or 5.0 mg capsule once daily (o.d) depending on previous treatment with RAAS blockers and up-titrated to ramipril 10 mg capsule o.d by end of period 1.
  In double blind phase (Period 2), patients received ramipril 10 mg capsule o.d and matching placebo of aliskiren tablet.
  Interventions: Drug: ramipril; Drug: Placebo to aliskiren
- Aliskiren plus Ramipril (Experimental): In open label run-in phase (period 1), patients started with ramipril 2.5 mg or 5.0 mg capsule once daily (o.d) depending on previous treatment with RAAS blockers and up-titrated to ramipril 10 mg capsule o.d by end of period 1.
  In double blind phase (period 2), patients received ramipril (10 mg once daily capsule) and aliskiren (150 mg once daily tablet) up titrated to 300 mg once daily after 1 week of treatment following a clinical safety patient assessment at the study site
  Interventions: Drug: aliskiren; Drug: ramipril

INTERVENTIONS:
Drug: aliskiren — Aliskiren 150 mg once daily up titrated to 300 mg once daily after 1 week of treatment following a clinical safety patient assessment at the study site
  Arms: Aliskiren; Aliskiren plus Ramipril
Drug: ramipril — 2.5 mg , 5.0 mg or 10 mg once daily
Drug: Placebo to aliskiren — matching placebo to aliskiren in double blind phase
  Arms: Ramipril
Drug: Placebo to ramipril — Matching placebo to ramipril capsule in double blind phase
  Arms: Aliskiren

SUMMARY:
In addition to the blood pressure lowering effects of aliskiren, it may have beneficial effects on blocking the so called RAAS (renin-angiotensin-aldosterone system) at the tissue level. An increase of angiotensin II is associated with progression of heart failure. Although the use of ACE-inhibitors in heart failure shows clinical benefit, an increase in angiotensin II due to an angiotensin II "escape" phenomenon is not desirable. It is not yet known if a direct renin inhibitor can reduce or even prevent the angiotensin II escape phenomenon associated with the use of an ACE-inhibitor. Therefore the study tested the effects of ramipril, aliskiren and the combination of both on levels of angiotensin II in the blood in patients with systolic heart failure

ELIGIBILITY:
Inclusion Criteria:

* Decompensated systolic heart failure, left ventricular ejection fraction ≤40%
* Brain natriuretic peptide (BNP) level ≥ 100 pg/mL

Exclusion criteria:

* Use of Angiotensin Converting Enzyme(ACE) or Angiotensin Receptor Blocker (ARB) inhibitor treatment following the run-in period or requirement of both treatments
* Acute heart failure secondary to acute myocardial infarction, acute coronary syndrome or new tachyarrhythmia
* Occurrence of unstable angina or myocardial infarction within 12 weeks prior to screening
* History of cardiomyopathy such as postpartum, restrictive, infective, hypertrophic obstructive
* History of right heart failure due to pulmonary disease
* History of untreated second or third degree atrioventricular heart block

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Germany (5):
  - Novartis Investigator Site, Bad Krozingen
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Göttingen
  - Novartis Investigator Site, Jena
  - Novartis Investigator Site, München
- Poland (5):
  - Novartis Investigator Site, Krakow
  - Novartis Investigator Site, Lublin
  - Novartis Investigator Site, Poznan
  - Novartis Investigator Site, Warsaw
  - Novartis Investigator Site, Wroclaw
- Russia (2):
  - Novartis Investigator Site, Moscow
  - Novartis Investigative Site, Moscow

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient enrolled to 4 week open label run-in phase (period 1) to up-titrate ramipril dose. 123 patients were randomized on Day 1 of Period 2 in a double-blind fashion to one of the three (1:1:1) treatment arms. The double-blind period was for 12 weeks.
Period: Overall Study
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Started | 40 ("Started" indicates randomized, safety and pharmacodynamic population) | 42 | 41
Completed | 40 | 38 | 38
Not Completed | 0 | 4 | 3
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Abnormal laboratory values | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril | Total
Number analyzed (Participants) | 40 | 42 | 41 | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.00) | 64.3 (9.91) | 62.0 (10.47) | 62.6 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 7 | 26
  Male | 29 | 34 | 34 | 97

OUTCOME MEASURES:

1. Primary Outcome: Venous Angiotensin II Levels After 12 Weeks of Treatment
Description: Peripheral venous blood was collected after 30 minutes of rest in the sitting position for analysis of biomarkers. Geometric mean ratio to baseline at Week 12 for Venous angiotensin II levels was calculated in patients with decompensated systolic heart failure (SHF) and left ventricular ejection fraction ≤40% at 0 hour pre-dose, 3 hours and 24 hours post-dose.
Time Frame: Baseline. 12 Weeks (Day 84, period 2)
Population: Pharmacodynamic (PD) Analysis Set: Subjects with any available PD data and no major protocol deviations with impact on PD data. Only patients with a value at both baseline and post-dose are included. In each category "n" indicates patients with observations at that time point.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Number analyzed (Participants) | 40 | 42 | 41
ratio
  0 Hour pre-dose (n=40, 38, 37) | 0.91 [0.52 to 1.59] | 1.08 [0.64 to 1.81] | 0.66 [0.37 to 1.18]
  3 hour post-dose (n=40, 38, 38) | 0.38 [0.23 to 0.62] | 0.44 [0.24 to 0.78] | 0.38 [0.22 to 0.66]
  24 hour post-dose (n=40, 38, 38) | 0.79 [0.44 to 1.41] | 0.97 [0.59 to 1.60] | 0.64 [0.34 to 1.24]

2. Secondary Outcome: Biomarker Plasma Renin Concentration (PRC)After 12 Weeks of Treatment
Description: Peripheral venous blood was collected after 30 minutes of rest in the sitting position for analysis of biomarkers. Geometric Mean Ratio to baseline at 12 weeks for PRC was calculated at 0 hour pre-dose.
Time Frame: Baseline, 12 weeks (84 days, period 2)
Population: Pharmacodynamic (PD) Analysis Set: Subjects with any available PD data and no major protocol deviations with impact on PD data. Only patients with a value at both baseline and post-dose are included.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Number analyzed (Participants) | 40 | 38 | 37
ratio | 2.48 [1.67 to 3.66] | 0.96 [0.71 to 1.30] | 4.67 [2.80 to 7.78]

3. Secondary Outcome: Biomarker Trapping Plasma Renin Activity (tPRA) After 12 Weeks of Treatment
Description: Peripheral venous blood was collected after 30 minutes of rest in the sitting position for analysis of biomarkers. Geometric Mean Ratio to baseline at Week 12 for tPRA was calculated at 0 hour pre-dose, 3 hour and 24 hour post-dose.
Time Frame: Baseline,12 weeks (84 days, Period 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Number analyzed (Participants) | 40 | 42 | 41
ratio
  0 hour pre-dose (n=40,38,37) | 0.14 [0.08 to 0.24] | 1.02 [0.68 to 1.52] | 0.25 [0.15 to 0.41]
  3 hour post-dose (n=40,38,38) | 0.07 [0.04 to 0.14] | 1.50 [0.86 to 2.61] | 0.15 [0.09 to 0.24]
  24 hour post-dose (n=40,38,38) | 0.12 [0.07 to 0.22] | 0.90 [0.58 to 1.40] | 0.16 [0.11 to 0.25]

4. Secondary Outcome: Biomarker B-type Natriuretic Peptide (BNP) After 12 Weeks of Treatment
Description: Peripheral venous blood was collected after 30 minutes of rest in the sitting position for analysis of biomarkers. Geometric Mean Ratio to baseline at Week 12 for BNP was calculated at 0 hours pre-dose.
Time Frame: Baseline, 12 weeks (Day 84 period 2)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Number analyzed (Participants) | 40 | 38 | 37
ratio | 0.96 [0.80 to 1.16] | 0.84 [0.69 to 1.03] | 0.78 [0.64 to 0.95]

5. Secondary Outcome: Biomarker Urinary Aldosterone After 12 Weeks of Treatment
Description: 24 hour urine collections were performed. Geometric Mean Ratio to baseline at Week 12 for Urinary aldosterone was calculated 24 hours post-dose.
Time Frame: Baseline,12 weeks (Day 84 period 2)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Ramipril | Aliskiren Plus Ramipril
Number analyzed (Participants) | 40 | 37 | 36
ratio | 0.83 [0.64 to 1.08] | 0.96 [0.78 to 1.18] | 0.87 [0.63 to 1.21]

6. Secondary Outcome: Pharmacokinetic of Aliskiren: Time to Reach the Maximum Concentration (Tmax) After Drug Administration
Description: Blood samples (2 mL) for the determination of aliskiren concentration in plasma were collected using an indwelling cannula inserted in a forearm vein. Samples were collected at week 12 (day 84): pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose.
Time Frame: 12 weeks
Population: All subjects with evaluable PK parameter data and no major protocol deviations with impact on PK data were included in the PK data analysis.
Measure: Median (Full Range); unit: Hour
Arm/Group | Aliskiren
Number analyzed (Participants) | 40
Hour | 1.50 (1.7896) [0.42 to 7.97]

7. Secondary Outcome: Pharmacokinetic of Aliskiren: The Observed Maximum Plasma Concentration (Cmax) Following Drug Administration
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aliskiren
Number analyzed (Participants) | 40
ng/mL | 257.2 (270.23)

8. Secondary Outcome: Pharmacokinetic of Aliskiren: The Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau(AUCtau)
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Aliskiren
Number analyzed (Participants) | 40
hr*ng/mL | 1707 (1321.9)

9. Secondary Outcome: Pharmacokinetic of Aliskiren: The Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast)
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Aliskiren
Number analyzed (Participants) | 40
hr*ng/mL | 3041 (1669.1)

10. Secondary Outcome: Pharmacokinetic of Aliskiren: The Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
hr*ng/mL | 3502 (1907.5)

11. Secondary Outcome: Pharmacokinetic of Aliskiren: The Terminal Elimination Half-life (T½)
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
hour | 31.02 (10.624)

ADVERSE EVENTS:
Description: Reported adverse events summarized events of the run-in period and double blind period. All serious adverse (SAEs) events were not suspected to be related to study drug
Groups:
- Ramipril + Aliskiren: In open label run-in phase (period 1), patients started with ramipril 2.5 mg or 5.0 mg capsule once daily (o.d) depending on previous treatment with RAAS blockers and up-titrated to ramipril 10 mg capsule o.d by end of period 1.
  In double blind phase (period 2), patients received ramipril (10 mg once daily capsule) and aliskiren (150 mg once daily tablet) up titrated to 300 mg once daily after 1 week of treatment following a clinical safety patient assessment at the study site.
Arm/Group | Ramipril | Aliskiren | Ramipril + Aliskiren
Serious Adverse Events (participants affected / at risk) | 7/42 | 2/40 | 3/41
Other Adverse Events (participants affected / at risk) | 6/42 | 3/40 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (N=42) | Aliskiren (N=40) | Ramipril + Aliskiren (N=41)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Sudden death (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (N=42) | Aliskiren (N=40) | Ramipril + Aliskiren (N=41)
Tachycardia (Cardiac disorders) | 0 | 1 | 5
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.